CLINICAL TRIAL: NCT06272812
Title: A Phase 2b, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy, Safety and Immunogenicity of a Candidate Tuberculosis (TB) Vaccine, MTBVAC, Against TB Disease in Interferon Gamma Release Assay Positive Adolescents and Adults Aged 14-45 Years, Living in a TB Endemic Region.
Brief Title: A Study to Evaluate the Efficacy, Safety and Immunogenicity of MTBVAC in IGRA Positive Adolescents and Adults Living in a TB Endemic Region.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Biofabri, SLU (Unknown); Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI C113
Record Dates: First submitted 2024-02-09; First posted 2024-02-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis (TB)
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTBVAC (Experimental): MTBVAC
  Interventions: Biological: MTBVAC
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MTBVAC — Vaccine Dose: MTBVAC 5x10^5 Formulation (approximately, per standard dose): 3 - 17x10^5 CFU Sucrose Sodium glutamate Presentation: Lyophilized pellet in vials (10 doses) Volume: 0.1 mL/dose Intradermal
  Arms: MTBVAC
Biological: Placebo — 0.9% saline Volume: 0.1 mL/dose Intradermal
  Arms: Placebo

SUMMARY:
A Phase 2b, double-blind, randomized, placebo-controlled study to evaluate the efficacy, safety and immunogenicity of a candidate tuberculosis (TB) vaccine, MTBVAC, against TB disease in interferon gamma release assay positive adolescents and adults aged 14-45 years, living in a TB endemic region.

DETAILED DESCRIPTION:
Phase 2b, double-blind, randomized, placebo-controlled, safety and efficacy study in 4,300 healthy adults and with a positive interferon gamma release assay (IGRA) test result. Most participants are likely to have received previous BCG vaccination in infancy. The investigational product is MTBVAC administered intradermally at 5x10^5 CFU.

Participants meeting the enrolment criteria will be randomized in a 1:1 ratio to receive a single dose of MTBVAC or placebo administered intradermally on Study Day 1.

Participants will be followed up for efficacy following vaccination via regular visits and contacts to screen for possible TB. Participants will also be trained to recognize signs and symptoms consistent with pulmonary TB disease and to report them for clinical evaluation. Participants with clinical presumption of pulmonary TB will be assessed with confirmatory diagnostic testing using a Nucleic Acid Amplification Test (Xpert MTB/RIF Ultra assay) and microbiological culture in sputum sampled on 3 separate days within a 1-week period. Participants diagnosed with pulmonary TB will be referred for TB treatment according to local clinical practice.

Only HIV-negative participants will be eligible for enrolment. Participants will be tested for HIV seroconversion at the end of each year of follow-up and at the presumptive TB visits. Participants who test positive for HIV will be referred for TB preventive treatment and antiretroviral treatment according to local clinical practice.

A sub-cohort of approximately 640 participants (320 in each study arm) will be selected for follow-up for solicited adverse events (AE) and selected chemistry and complete blood count (CBC). Additionally, a sub-cohort of approximately 430 participants (215 in each study arm) will be selected for specific immunogenicity assessments. The strategy for participant sub-cohort selection will be described in the Study Operations Manual (SOM).

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged 14 through 45 years on Study Day 1.
2. Has completed the written (or thumb printed and witnessed) informed consent process (participants older than 18 years) or has completed the written parental consent and participant assent process (participants younger than 18 years) before any study-related procedures were performed.
3. Participants who, in the opinion of the investigatory, can and will comply with the requirements of the protocol (e.g., to stay in contact with the Clinical Research Centre (CRC), return for follow-up visits)
4. Has general good health as confirmed by medical history and physical examination.
5. All participants born female who are engaging in sexual activity that could lead to pregnancy must commit to use an acceptable method of contraception from 21 days prior to Study Day 1 and for the 2 months after vaccination. Acceptable contraception includes:

   1. Condoms (male or female) with or without spermicide
   2. Diaphragm or cervical cap with spermicide
   3. Intrauterine device
   4. Hormonal contraception (combined estrogen and progestogen, or progestogen-only), including contraceptive implant or injectable
   5. Successful vasectomy in the male partner, considered successful if a woman reports that a male partner has:

      documentation of azoospermia by microscopy (1 year ago) or a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy
   6. Not of reproductive potential, such as having undergone hysterectomy, bilateral oophorectomy or tubal ligation, postmenopausal (any age and amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 IU/L), surgically sterile.
   7. Sexual abstinence. All participants born female who are not heterosexually active at screening must agree to utilize an acceptable method of contraception if they become heterosexually active as outlined above.
6. All male participants should agree to use barrier contraception with their female partners for at least 2 weeks after vaccination.
7. Has not shared the same enclosed living space with someone diagnosed with TB for one or more nights or for frequent or extended daytime periods during the 6 months prior to Study Day 1.
8. Has a positive IGRA test result at screening.
9. HIV negative at screening.
10. Negative clinical screening questionnaire and Xpert MTB/RIF negative sputum sample for pulmonary TB disease at screening.

Exclusion Criteria:

1. Acute illness and/or axillary temperature ≥37.5°C on Study Day 1.
2. Current suspicion or evidence (including but not limited to sputum Xpert MTB/RIF positive) of active TB disease at any CRC. An attempt must be made to obtain sputum from each participant; persons who are sputum unproductive will be assumed to be Xpert MTB/RIF negative.
3. History of previous TB disease and/or treatment for TB disease.
4. History of TB preventative therapy, not including BCG vaccination.
5. Received any investigational drug or investigational vaccine within 42 days before Study Day 1, or planned use during the study period.
6. Planned administration/administration of a licensed vaccine not foreseen by the study protocol in the period starting 28 days before Study Day 1 and ending 28 days after vaccine administration.
7. Prior receipt of any investigational TB vaccine candidate before Study Day 1. Note: receipt of placebo in a previous TB vaccine trial will not exclude a participant from participation if documentation is available and the Medical Monitor gives approval.
8. Chronic administration of immunosuppressive medication within 42 days before Study Day 1 (inhaled and topical corticosteroids are permitted).
9. Any confirmed or suspected immunosuppressive, immunodeficient, or autoimmune condition based on medical history and physical examination (no laboratory testing required).
10. Concurrent, or planned participation in any other investigational study during the study period. (Concurrent participation in an observational trial not requiring blood or tissue sample collection is not an exclusion.)
11. Received immunoglobulin or blood products within 42 days before Study Day 1, or planned administration during the study period.
12. History or any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
13. Pregnant or lactating/nursing female, or positive urine pregnancy test during screening or pre-vaccination on Study Day 1.
14. Any current, or history of, medication use or medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, might compromise the safety of the participant or make it unlikely that the participant will comply with the protocol.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4300 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the protective efficacy of of MTBVAC against bacteriologically confirmed pulmonary TB disease, diagnosed by more than one diagnostic test with sputum obtained before initiation of TB treatment as compared to placebo. | 36 Months
  Incident cases of definite pulmonary TB disease in participants with clinical suspicion of pulmonary TB disease, with Mtb identified by at least two positive diagnostic tests (microbiological culture, Xpert MTB/RIF Ultra, or both) from sputum specimens taken before initiation of TB treatment and confirmed HIV-negative at the time of TB diagnosis, over a period starting 28 days following vaccination and lasting up to 36 months post vaccination.

SECONDARY OUTCOMES:
To evaluate the protective efficacy of one dose of MTBVAC against bacteriologically confirmed pulmonary TB disease, not associated with HIV infection, diagnosed with sputum obtained before initiation of TB treatment, as compared to placebo. | 36 Months
  Incident cases of definite pulmonary TB disease in participants with clinical suspicion of pulmonary TB disease, with Mtb identified by microbiological culture and/or Xpert MTB/RIF Ultra from sputum specimens taken before initiation of TB treatment and confirmed HIV-negative at the time of TB diagnosis, over a period starting 28 days following vaccination and lasting up to 36 months post vaccination.
To evaluate the protective efficacy of MTBVAC candidate vaccine against definite Xpert MTB/RIF Ultra positive pulmonary TB disease diagnosed with sputum obtained before initiation of TB treatment, as compared to placebo. | 36 months
  Incident cases of definite pulmonary TB disease in participants with clinical suspicion of pulmonary TB disease, with Mtb identified by Xpert MTB/RIF Ultra from sputum specimens taken before initiation of TB treatment and confirmed HIV-negative at the time of TB diagnosis, over a period starting 28 days following vaccination and lasting up to 36 months post last vaccination.
To evaluate the protective efficacy of one dose of MTBVAC candidate vaccine against clinical TB, as compared to placebo | 36 months
  Incident cases of clinical TB disease diagnosed by a clinician who has decided to treat the patient with TB treatment, over a period starting 28 days following vaccination and lasting up to 36 months post last vaccination
To assess the safety and reactogenicity of one dose of MTBVAC candidate vaccine. | 6 Months
  Occurrence of all SAEs until Month 6 following vaccination.
To assess the safety and reactogenicity of one dose of MTBVAC candidate vaccine. | 36 months
  Occurrence of vaccine related SAEs during the entire study period.
To assess the safety and reactogenicity of one dose of MTBVAC candidate vaccine. | 7 Days
  Occurrence of solicited local and systemic AEs in the safety sub-cohort during the 7 days following vaccination (day of vaccination and 6 subsequent days).
To assess the safety and reactogenicity of one dose of MTBVAC candidate vaccine. | 28 Days
  Occurrence of unsolicited AEs during the 28 days following vaccination (day of vaccination and 27 subsequent days).
To assess the safety and reactogenicity of one dose of MTBVAC candidate vaccine. | 84 Days
  Occurrence of grade 3 or higher injection site reactions during the 84 days following vaccination (day of vaccination and 84 subsequent days).
To assess the safety and reactogenicity of one dose of MTBVAC candidate vaccine. | 36 months
  Occurrence of grade 2 or higher haematological and chemistry abnormalities, in the safety sub-cohort.
To assess the immunogenicity of one dose of the MTBVAC candidate vaccine via assessment of humoral and cell-mediated immune (CMI) responses in a subset of the enrolled participants. | 36 months
  Evaluation of CMI responses with respect to components of the study vaccine, in the immunogenicity sub-cohort at Day 1 (prior to vaccination), Day 29, Month 12, Month 24 and Month 36 (if applicable).
To assess the immunogenicity of one dose of the MTBVAC candidate vaccine via assessment of humoral and cell-mediated immune (CMI) responses in a subset of the enrolled participants. | 36 months
  Evaluation of humoral immune responses with respect to components of the study vaccine, in the immunogenicity sub-cohort at Day 1 (prior to vaccination), Day 29, Month 12, Month 24 and Month 36 (if applicable).

CONTACTS AND LOCATIONS:
Locations (1):
- The Aurum Institute Tembisa Clinical Research Centre, Johannesburg, South Africa